CLINICAL TRIAL: NCT07324824
Title: Sintilimab Combined With Bevacizumab as Neoadjuvant Therapy for Resectable Hepatocellular Carcinoma Beyond the Milan Criteria: A Single-Arm, Prospective Phase II Study
Brief Title: Sintilimab Plus Bevacizumab Biosimilar as Neoadjuvant Therapy for Resectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-720-01
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; Neoadjuvant Therapy; Sintilimab; Bevacizimab
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sintilimab combined with bevacizumab biosimilar (Experimental)
  Interventions: Drug: sintilimab combined with bevacizumab biosimilar

INTERVENTIONS:
Drug: sintilimab combined with bevacizumab biosimilar — Drug: Sintilimab: 200mg IV Q3W D1 (3 cycles) Drug: Bevacizumab Biosimilar: 15mg/kg, IV, Q3W, D1 (2 cycles)

SUMMARY:
Surgical resection is the preferred therapeutic modality for patients with resectable hepatocellular carcinoma (HCC). However, the recurrence rate of HCC remains up to 70%. Neoadjuvant therapy for HCC could potentially reduce the risk of postoperative recurrence and prolong overall survival. Nevertheless, there is no standard neoadjuvant treatment regimen for HCC to date. In recent years, targeted therapy and immunotherapy are proved to improve the prognosis of advanced HCC patients. Previous study (ORIENT-32) has confirmed that, compared with sorafenib, sintilimab combined with bevacizumab biosimilar can delay tumor progression, reduce the risk of death, and exhibit a favorable safety profile in patients with advanced HCC. Therefore, we conducted a prospective, single-arm phase II study to investigate the efficacy of sintilimab combined with a bevacizumab biosimilar as neoadjuvant therapy in patients with resectable HCC beyond the Milan criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent and willing to sign an approved consent form;
2. Aged ≥ 18 years;
3. Clinically diagnosed or pathologically confirmed resectable hepatocellular carcinoma beyond the Milan criteria (CNLC Ib-IIa);
4. No prior anti-HCC treatment;
5. Child-Pugh class A.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
7. Expected survival time of > 6 months.
8. Sufficient organ and bone marrow function.

Exclusion Criteria:

1. Known as cholangiocarcinoma (ICC) or mixed hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and hepatic fibrolamellar carcinoma;
2. History of organ transplantation or hepatic encephalopathy
3. Pleural fluid, ascites, and pericardial effusion with clinical symptoms requiring drainage
4. History of esophageal or gastric variceal bleeding caused by portal hypertension within the past 6 months; Documented severe (Grade 3) varices identified by endoscopy within 3 months prior to enrollment; Evidence of portal hypertension and assessed by the investigator as being at high risk of bleeding.
5. Arterial and venous thromboembolic events in the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or any other serious thromboembolism history;
6. Any life-threatening bleeding event occurring within the past 3 months;
7. Severe bleeding tendency, coagulopathy, or ongoing thrombolytic therapy.
8. Chronic requirement for medications that inhibit platelet function, such as aspirin (>325 mg/day), dipyridamole, or clopidogrel.
9. Uncontrolled hypertension, defined as systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg despite optimal medical management; history of hypertensive crisis or hypertensive encephalopathy.
10. Symptomatic congestive heart failure (New York Heart Association [NYHA] Functional Class II-IV); symptomatic or poorly controlled arrhythmias; history of congenital long QT syndrome; or corrected QT interval (QTc) >500 ms at screening (calculated using Fridericia's formula).
11. History of gastrointestinal perforation and/or fistula, intestinal obstruction (including incomplete obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection complicated by chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic persistent diarrhea within the past 6 months.
12. Major surgical procedure (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to enrollment; presence of unhealed wounds, ulcers, or fractures; or tissue biopsy or other minor surgical procedure within 7 days prior to enrollment, excluding venous catheterization for intravenous infusion.
13. Past or current history of pulmonary diseases including pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-induced pneumonia, or severe impairment of lung function.
14. Active acute or chronic hepatitis B or C infection, defined as: hepatitis B virus (HBV) DNA >2000 IU/mL or 10⁴ copies/mL; hepatitis C virus (HCV) RNA >10³ copies/mL; or concurrent positivity for hepatitis B surface antigen (HBsAg) and anti-HCV antibodies.
15. Active tuberculosis (TB); ongoing anti-TB treatment; or anti-TB treatment completed within 1 year prior to the initiation of study treatment.
16. Human immunodeficiency virus (HIV) infection (positive for HIV 1/2 antibodies); known syphilis infection.
17. Severe active infection or infection with poor clinical control.
18. Active autoimmune disease requiring systemic therapy (e.g., disease-modifying antirheumatic drugs, corticosteroids, or immunosuppressants) within 2 years prior to enrollment. Substitution therapy (e.g., thyroid hormone, insulin, or physiological doses of corticosteroids for adrenal or pituitary insufficiency) is permitted. A history of known primary immunodeficiency is excluded. Patients with isolated positive autoimmune antibodies must be evaluated by the investigator to confirm the absence of underlying autoimmune disease.
19. Use of immunosuppressive drugs within 4 weeks prior to enrollment, excluding intranasal, inhaled, or other topical corticosteroids, or systemic corticosteroids at physiological doses (i.e., ≤10 mg/day of prednisone or equivalent). Temporary use of corticosteroids for the management of dyspnea related to asthma, chronic obstructive pulmonary disease (COPD), or other conditions is permitted.
20. Administration of live-attenuated vaccines within 4 weeks prior to enrollment or planned administration of live-attenuated vaccines during the study period.
21. Use of immunomodulatory agents (including thymosin, interferons, or interleukins) within 2 weeks prior to enrollment, excluding local administration for the control of pleural effusion or ascites.
22. Uncontrolled/uncorrectable metabolic disorders, other non-malignant organ/systemic diseases, or cancer-related sequelae that pose a high medical risk and/or introduce uncertainty in survival assessment.
23. Diagnosis of other malignant tumors within 5 years prior to enrollment, excluding curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or curatively resected carcinoma in situ. For malignant tumors diagnosed more than 5 years prior to drug administration, pathological or cytological confirmation of recurrent or metastatic lesions is required.
24. Prior receipt of any anti-angiogenic agents, anti-PD-1 antibodies, anti-PD-L1/L2 antibodies, anti-CTLA-4 antibodies, or other immunotherapies.
25. Known hypersensitivity to sintilimab, bevacizumab formulations, or their excipients; or history of severe hypersensitivity reactions to other monoclonal antibodies.
26. Receipt of treatment in other clinical trials within 4 weeks prior to enrollment.
27. Pregnant or breastfeeding female patients.
28. Other acute or chronic diseases, psychiatric disorders, or abnormal laboratory findings that, in the investigator's judgment, would: increase the risk associated with study participation or study drug administration; interfere with the interpretation of study results; or render the patient ineligible for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence free survival rate | Up to 2 years
  Defined as the proportion of patients who remain free from any tumor recurrence or death within 1 year after liver resection.
Adverse Events (AEs) | Up to 2 years
  Defined as the proportion of patients with AEs assessed by NCI CTCAE v5.0;

SECONDARY OUTCOMES:
R0 resection rate | Up to 2 years
  Defined as the proportion of patients received R0 resection
pathological complete response | Up to 2 years
  Defined as the proportion of patients who had pathological complete response
major pathological response | Up to 2 years
  Defined as the proportion of patients who had major pathological response
Overall survival | Up to 2 years
  Defined as the interval from the date of enrollment to the date of death or to the date of last follow-up (whichever occurs first)
Recurrence free survival | Up to 2 years
  Defined as the time from the date of liver resection to the date of recurrence or death (whichever occurs first)
Time to recurrence | Up to 2 years
  Defined as the time from the date of liver resection to the date of tumor recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided